CLINICAL TRIAL: NCT03611569
Title: Interventional, Randomized, Double-blind, Sequential-group, Placebo-controlled, Single-ascending-dose Study Investigating the Safety, Tolerability and Pharmacokinetic and Pharmacodynamic Properties of Lu AF82422 in Healthy Non-Japanese and Japanese Subjects and in Patients With Parkinson's Disease
Brief Title: Lu AF82422 in Healthy Non-Japanese and Japanese Subjects and in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 17699A
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Healthy; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Cohort
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AF82422 (Experimental): Part A:
  Cohort A1, A2, and A3: 24 healthy subjects, with 8 subjects per cohort (aiming for an equal number of men and women) Cohort A4,A5,A6: 36 healthy subjects, with 6 non-Japanese subjects and 6 Japanese subjects per cohort (aiming for an equal number of men and women)
  Part B:
  Cohort B1, B2, B3: 24 patients with Parkinson's disease
  Interventions: Drug: Lu AF82422
- Placebo (Placebo Comparator): Part A:
  Cohort A1, A2, and A3: 24 healthy subjects, with 8 subjects per cohort (aiming for an equal number of men and women) Cohort A4,A5,A6: 36 healthy subjects, with 6 non-Japanese subjects and 6 Japanese subjects per cohort (aiming for an equal number of men and women)
  Part B:
  Cohort B1, B2, B3: 24 patients with Parkinson's disease
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AF82422 — Lu AF82422 - concentrate for solution for infusion; vials containing 50mg/ml, single dose
  Arms: Lu AF82422
Drug: Placebo — placebo - concentrate for solution for infusion, single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety of a single dose of Lu AF82422, how well it is tolerated, how the drug effects the body and what the body does to the drug in healthy non-Japanese and Japanese subjects and in patients with Parkinson's disease

ELIGIBILITY:
Inclusion criteria:

Healthy subjects:

- Men and women ≥18 and ≤55 years of age with a body mass index (BMI) ≥18 and ≤32 kg/m2 (non-Japanese subjects) and ≥18 and ≤28 kg/m2 (Japanese subjects)

Patients with Parkinson's disease:

* Men and women with a clinical diagnosis of idiopathic Parkinson's disease, Hoehn and Yahn (H&Y, stage 1-3)
* For a minimum of three months prior to enrolment, Parkinson's disease symptoms have been stable and is anticipated to be stable during the study duration as judged by the PI
* If on Parkinson's disease treatment the dose must be stable for a minimum of three months prior to enrolment and is anticipated to be stable during the study duration as judged by the PI
* ≥40 and ≤80 years of age
* BMI ≥18 and ≤35 kg/m2

Exclusion criteria:

* Atypical Parkinsonism
* Clinically relevant structural brain abnormality, as assessed using MRI
* Mild cognitive impairment, measured as a Montreal cognitive assessment (MoCA) score =<21
* Any past or current treatment with an active vaccine targeting alpha-synuclein
* Any past or current treatment with a monoclonal antibody within the last 12 months

Other in- and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From dosing to Day 84
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, blood closure time and ECG parameters)

SECONDARY OUTCOMES:
AUC 0-t | From dosing to Day 84
  Area under the Lu AF82422 plasma concentration curve from zero to time t
Cmax | From dosing to Day 84
  Maximum observed plasma concentration of Lu AF82422
CL | From dosing to Day 84
  Clearance of Lu AF82422

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (4):
- United States (4):
  - California Clinical Trials Medical Group (CCTMG), Glendale, California
  - Reserach Center of America, Hollywood, Florida
  - PPD, Orlando, Florida
  - Parexel, Early Phase Clinical Unit (EPCU), Harbor Hospital, Baltimore, Maryland